CLINICAL TRIAL: NCT01424956
Title: To Determine the Impact on Reader Performance, as Defined by the Area Under the Receiver Operating Characteristic Curve, When Automated Breast Ultrasound and a Screening Mammogram Are Combined, Compared to a Screening Mammogram Alone in Asymptomatic Women With >50% Parenchymal Density and a Screening Mammogram Assigned a BI-RADS Assessment Category 1 (Negative) or 2 (Normal With Benign Findings).
Brief Title: CRRS-4 Pivotal Somo•v™ ABUS ROC Reader Observer Study
Status: Completed | Type: Observational
Sponsor: U-Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: USI2011001
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
Keywords: breast; breast cancer; breast screening; breast cancer screening; ultrasound; ultrasonography; mammogram; mammography; breast density; dense breasts; early detection; somo v; somo•v; U-Systems; Automated Breast Ultrasound; Ultrasonography, Mammary; Breast Neoplasms; Breast Density > 50% (BI-RADS III & IV)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asymptomatic Women who have Dense Breast Tissue: Women who have no signs or symptoms of breast cancer who have > 50% parenchymal density on mammography.
  Interventions: Device: Automated Breast Ultrasound (ABUS)

INTERVENTIONS:
Device: Automated Breast Ultrasound (ABUS) — Automated Breast Ultrasound (ABUS) as an adjunct to digital screening mammography.
  Other Names: somo.V ABUS; ABUS; Whole Breast Ultrasound

SUMMARY:
To determine the impact on Interpreting Physician performance in detecting breast cancer, as defined by the area under the Receiver Operating Characteristic Curve (ROC), when Automated Breast Ultrasound (ABUS) and screening mammography (XRM) are combined, compared to screening mammography alone in asymptomatic women with >50% parenchymal density and a screening mammogram assigned a BI-RADS Assessment Category 1 (negative) or 2 (normal with benign findings).

The effect of the improved Reader performance is illustrated by plotting the ROC curves for XRM alone and XRM+ABUS. If Reader performance improves with the addition of ABUS to the XRM, the area under the curve (AUC) for XRM+ABUS (AUCXRM+ABUS) will be greater than the area under the curve for XRM Alone (AUCXRM Alone). This difference is represented as ∆AUCABUS. The null and alternative hypotheses can be formally expressed as follows:

H0: ∆AUCABUS = 0, AUCXRM+ABUS = AUCXRM Alone The null hypothesis is that Reader performance will be unchanged with the addition of ABUS to a screening mammogram assigned a BI-RADS Assessment Category of 1 or 2.

HA: ∆AUCABUS ≠ 0, AUCXRM+ABUS ≠ AUCXRM Alone The alternative hypothesis is that Reader performance will be changed with the addition of ABUS to a screening mammogram assigned a BI-RADS Assessment Category of 1 or 2. A statistically significant change will be considered equivalent to a statistically significant improvement if the estimated value of AUCXRM+ABUS is greater than that of AUCXRM Alone with statistical significance at an alpha level of .05 for a two-sided test.

DETAILED DESCRIPTION:
The Clinical Retrospective Reader Study is an observational case-controlled, multi-reader multi-case Receiver Operating Characteristic (ROC) study involving approximately 16 Interpreting Physicians (Readers) and approximately 200 breast screening cases which will be reviewed and of those, 164 breast screening cases will be included in the primary data analysis. All primary data analysis cases will consist of screening mammogram and Automated Breast Ultrasound image readings from the same asymptomatic females with >50% parenchymal density for whom the screening mammogram was assigned a BI-RADS Assessment Category 1 (negative) or 2 (normal with benign findings).

The Readers will review a total of 200 cases: the Non-Cancer Case Set, the Cancer Case Set, and additional Control and Supplemental Case Sets. These cases will be randomized during the reading session so each Reader will review the entire Case Set in a unique order.

The primary Receiver Operating Characteristic analysis will be performed on the Readers' Likelihood of Malignancy (LOM) ratings from their initial review of the screening mammogram alone and their final review of the screening mammogram and Automated Breast Ultrasound for the Non-Cancer Case Set and Cancer Case Set.

ELIGIBILITY:
Inclusion Criteria:

* Interpreting Physician as defined under 21CFR §900.12(a)(1)(i)(B)(2).
* Fellowship-Trained in Breast Imaging and or have 10 years experience in breast imaging in which the radiologist's practice was at least 70% breast imaging
* Currently meets the minimum Mammography Interpretation requirements per MQSA
* Review Rate of at least 1,000 Mammograms annually for the year prior to study participation
* Review Rate of at least 500 Breast Ultrasounds annually for the year prior to study participation
* Successful completion of ABUS training

Exclusion Criteria:

* Does not meet definition of Interpreting Physician as defined under 21CFR §900.12(a)(1)(i)(B)(2).
* Does not meet requirements of Fellowship-Trained in Breast Imaging and or have 10 years experience in breast imaging in which the radiologist's practice was at least 70% breast imaging
* Does not meet requirements of minimum Mammography Interpretation requirements per MQSA
* Does not meet requirements of Review Rate of at least 1,000 Mammograms annually for the year prior to study participation
* Does not meet requirements of Review Rate of at least 500 Breast Ultrasounds annually for the year prior to study participation
* Does not meet requirements of successful completion of ABUS training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 17 Interpreting Physicians (Readers) qualified by training and experience, who are in breast imaging practices in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Interpreting Physician Performance In Detecting Breast Cancer | Two months
  To determine the impact on Interpreting Physician (Reader) Performance in detecting breast cancer, as defined by the area under the Receiver Operating Characteristic (ROC) Curve (AUC), when ABUS and XRM are combined (XRM+ABUS), compared to XRM Alone in asymptomatic women with >50% parenchymal density (BI-RADS Composition/Density rating of 3 or 4) and a screening mammogram assigned a BI-RADS Assessment Category 1 (negative) or 2 (normal with benign findings).

SECONDARY OUTCOMES:
Interpreting Physician sensitivity and specificity of breast cancer detection. | Two months
  Reader sensitivity and specificity when XRM+ABUS are combined compared to XRM Alone for two different combinations of cut points.

CONTACTS AND LOCATIONS:
Overall Officials: Maryellen Giger, Ph.D., Principal Investigator — University of Chicago, Department of Radiology
Locations (1):
- U-Systems, Inc., Sunnyvale, California, United States